CLINICAL TRIAL: NCT06119412
Title: An Alternative Technique for Measuring Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Evrim Eyikara, Doctor Research assistant, Principal Investigator, Gazi University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: GaziU-SBF-EE-02
Record Dates: First submitted 2023-10-20; First posted 2023-11-07 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1, starting with standard technique (Other): According to block randomization, the 1st researcher will first apply the standard technique (60 seconds pause between palpation and auscultation), 1 minute break will be given, and the 2nd researcher will apply the alternative new technique (no break between palpation and auscultation) on the same person.
  Interventions: Other: blood pressure measurement starting with standard technique or alternative new technique. manual sphygmomanometer will be used.
- group 2, starting with alternative new technique (Other): According to block randomization, Investigator 1 will first apply the alternative new technique (no pause between palpation and auscultation) to the people in the second group, and a 1-minute break will be given. The 2nd researcher will apply the standard technique (60 seconds break between palpation and auscultation) on the same person.
  Interventions: Other: blood pressure measurement starting with standard technique or alternative new technique. manual sphygmomanometer will be used.

INTERVENTIONS:
Other: blood pressure measurement starting with standard technique or alternative new technique. manual sphygmomanometer will be used. — Each participant will have their blood pressure measured with two different techniques.

SUMMARY:
This cross design study will be conducted to evaluate the combination of palpation and auscultation techniques as an alternative technique for the measurement of blood pressure. The main questions it aims to answer are:

* Is there a statistical difference between the results of systolic blood pressure measured with the old and new technique?
* Is there a statistical difference between the results of systolic blood pressure measured with the old and new technique? Participants' blood pressure will be measured twice.

DETAILED DESCRIPTION:
As a result of clinical observations, a common practice is to inflate the cuff to a high and random mmHg value and start auscultation directly. Alternatively, many healthcare workers determine the moment when pulse beats disappear by palpation and increase this value by 30 mmHg without lowering the cuff and without taking a break for 1-2 minutes and start auscultation. In the literature, there is a similar technique called "one-step method". According to this technique, the sphygmomanometer is wrapped around the individual's arm and the stethoscope is placed in the ear. The brachial artery is then palpated and identified. The cuff is inflated up to 30 mmHg above the systolic blood pressure of the individual. The cuff is then depressurized to 2-3 mmHg/second. It is observed that many healthcare professionals and students use this technique today because it is more practical in terms of measurement time. However, it is thought that the step of "inflating the cuff up to 30 mmHg above the systolic blood pressure value of the individual" in the process steps of the technique is not reliable enough. It is thought that it may lead to erroneous results in capturing sudden blood pressure changes in the individual. In this context, it is thought that it would be more reliable to determine the value at the moment when the pulse is not felt with the palpation technique, add 30 mmHg to this value without interruption and without lowering the cuff and continue auscultation. At the same time, combining palpation and auscultation and continuing them consecutively will shorten the measurement time and provide a practical application.

It is aimed to measure blood pressure in approximately 202 healthy adults. The purpose and method of the study will be explained in detail to all participants included in the sample group. Participants will be allowed to rest for 15-30 minutes before blood pressure measurement. Blood pressure will be measured with two different techniques according to the order in which the participants are included in the study. The first participant's blood pressure will first be measured with the standard technique in the literature (with a break between palpation and auscultation). After a 60-second pause, blood pressure will be measured with the alternative recommended technique (palpation and auscultation combined). In the second participant, blood pressure will be measured first with the alternative recommended technique (combining palpation and auscultation). After a 60-second break and with the arm in the same position, blood pressure will be measured with the standard technique in the literature (with a break between palpation and auscultation). The cross-over method will be applied as possible differences between measurement times should be taken into account.

ELIGIBILITY:
Inclusion criteria:

* Over 18 years of age,
* no chronic disease,
* not taking any medication and/or treatment that affects the cardiovascular or circulatory system,
* volunteering to participate in the research.

Exclusion Criteria:

* has a chronic disease,
* taking medication that affects the cardiovascular or circulatory system,
* wants to leave the study at any stage.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
blood pressure measurement list | approximately 12 weeks from the start of measurements until reporting.
  This form will record the participant's systolic and diastolic blood pressure measured with the standard technique and the alternative new technique.

SECONDARY OUTCOMES:
blood pressure measurement time | approximately 12 weeks from the start of measurements until reporting.
  The number of seconds the blood pressure measurements last will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Eyikara, Principal Investigator — doctor research assistant
Locations (1):
- Gazi University Department of Health Sciences, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No